CLINICAL TRIAL: NCT07209280
Title: Cannulated Bone Bolt® Screw System Versus Standard Cannulated Screw System Fixation for Lateral Compression Type-1 (LC-1) Pelvic Ring Injuries: Multicenter Prospective Observational Study
Brief Title: Cannulated Bone Bolt® Screw System Versus Standard Cannulated Screw System Fixation for Pelvic Fractures
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lucas Marchand, Principle Investigator, University of Utah
Other Study IDs: 188952
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: Lateral Compression Type-1 (LC-1) fractures; Pelvic Ring Injuries; Cannulated Bone Bolt® Screw System; Standard Cannulated Screw System; Post-operative pain; Visual Analog Scale (VAS)
MeSH Terms: conditions — Pain; Fractures, Bone; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cannulated Bone Bolt® Screw System: Surgeons identifying as users of the Cannulated Bone Bolt® screws will be required to place at least one Cannulated Bone Bolt® screw in each of their operative LC1 injuries.
  Interventions: Other: Cannulated Bone Bolt® Screw System
- Standard Cannulated Screw System Fixation: Surgeons identifying as users of standard cannulated screws will be able to use the cannulated screw of their choice.
  Interventions: Other: Standard Cannulated Screw System

INTERVENTIONS:
Other: Cannulated Bone Bolt® Screw System — Patients treated with the Cannulated Bone Bolt® screw system for Lateral Compression Type -1 (LC-1) fractures.
  Groups: Cannulated Bone Bolt® Screw System
Other: Standard Cannulated Screw System — Patients treated with the Standard Cannulated Screw System for Lateral Compression Type -1 (LC-1) fractures.
  Groups: Standard Cannulated Screw System Fixation

SUMMARY:
The investigators aim is to determine if the cannulated Bone Bolt® screw system will provide improved post-operative pain control as compared to standard cannulated screw system fixation for the operative treatment of LC1 fractures (primary outcome). Hypothesis: Patients treated with the cannulated Bone Bolt® screw system will experience a clinically important difference (1.5 points) in post-operative pain as measured by the Visual Analog Scale (VAS) compared to patients treated with standard cannulated screw system fixation.

DETAILED DESCRIPTION:
Lateral Compression type-1 (LC1) fractures of the pelvis represent the most common injury to the pelvic ring, accounting for more than 50% of all pelvic ring injuries. These injuries occur secondary to a lateral compressive force on the pelvic ring causing an internal rotation force coupled with medialization of the impacted hemi-pelvis. Despite their prevalence, treatment algorithms for these injuries remain controversial. When significant deformity exists (>1cm displacement) the preference is typically for operative fixation as this has been listed repeatedly as an indication for surgery. In the setting of a minimally displaced LC1 fractures surgical indications become less clear. Minimally displaced fractures can have instability that is under appreciated on static imaging and can result in displacement with non-operative management. This has prompted many surgeons to treat the minimally displaced fracture more aggressively. Surgical intervention provides the benefit of preventing displacement, improving pain, and potentially progressing post-operative mobility.

Previous work has demonstrated short term benefit to the surgical treatment of these injuries, although the treatment benefits noted have been small. A recent observational study conducted at 16 trauma centers prospectively measured short-term VAS pain scores in 194 patients with unilateral sacral fractures and noted that patients with surgical fixation reported 2.7 points less pain at 24 hours postinjury (p=0.001) and 1.1 points less pain at 3 months as compared to those patients treated without surgery (p=0.02). Subsequent to this, an investigator demonstrated a small improvement in pain and functional outcome for up to 12 months in minimally displaced LC1 fractures with complete sacral injuries that were treated with surgical intervention as compared to those patients managed conservatively.

With this information at hand, the current treatment controversy for these injuries has shifted to determining how to optimize surgical fixation and pelvic stability, improve short-term outcomes such as pain, time to mobilization, discharge disposition, and physical function. Many surgeons now consider the short term benefits of surgical intervention to outweigh the risks of percutaneous pelvic fixation, and are desiring a more structurally reliable way in which surgical management to further improve consistency of patient outcomes. Present data provides little to no guidance as to which type of surgical fixation strategy may prove most beneficial to these patients and few advancements have been made in the technology used to treat pelvic ring injuries over the past several decades.

Standard treatment strategies for operative LC1 injuries includes management with cannulated sacroiliac (SI) or trans-sacral (TS) screws in the posterior pelvic ring with or without anterior pelvic ring fixation. Standard cannulated screw System fixation work reasonably well, but loosening and loss of fixation integrity are not infrequent. New advances in FDA cleared screw designs that offer greater mechanical stability, may give more reliable results from surgical treatment.

Given that improvements have been noted with surgical intervention but current surgical techniques and technology have only offered modest clinical benefits, the next logical step is to determine if new technology such as the Cannulated Bone Bolt® Screw System with proven increase mechanical strength and stiffness can improve post-operative patient outcomes. Given that these injuries represent the most common pelvic ring fractures but do not yet have a ideal and fully reliable treatment pathway, the results of this prospective study could greatly improve care of these patients. A prospective observational design is preferred given a true equipoise for screw design used in the operative treatments for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age at presentation between 18 and 80 years in line with literature from prior investigations.
* Operative LC1 pelvic ring injury.
* Glasgow Coma Scale of 15.
* Willingness to participate in study.

Exclusion Criteria:

* Inability to provide informed consent.
* Pregnant or lactating woman.
* Current incarceration.
* Associated spinal cord injury.
* Non-ambulatory patients (including patients with associated lower extremity fracture that may limit post-operative weight bearing).
* Patient presents with osteoporosis, which in the opinion of the Principal Investigator, may limit the subject's ability to support fracture repair using the study device.
* Patient has a metabolic disorder that may impair bone formation.
* Patient has osteomalacia.
* Patient has distant foci of infections which may spread to the implant site or patient with infection, sepsis or osteomyelitis.
* Patient has a vascular insufficiency, muscular atrophy, or neuromuscular disease.
* Patient is a current alcohol or drug abuser.
* Patients unable to comply with post-operative instruction.
* Other lower extremity injuries that impact weight bearing recommendation.
* Injuries that may have a larger impact on pain than the studied pelvic ring.
* Non-English/Spanish speaking.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 80 years with operative LC1 pelvic ring injury.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain | 2-weeks after surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 6-weeks after surgery
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 12-weeks after surgery
  VAS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Marchand, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No